CLINICAL TRIAL: NCT04076124
Title: Different Forms of Prefrontal Transcranial Stimulation and Brain-derived Neurotrophic Factor in the Prediction of Antidepressant Efficacy of Brain Stimulation
Brief Title: Brain-derived Neurotrophic Factor and the Antidepressant Efficacy of Brain Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: V107C-123
Record Dates: First submitted 2019-07-26; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active rTMS-DLPFC (Experimental): This active group will receive high-frequency repetitive TMS stimulation.
  Interventions: Device: Active rTMS-DLPFC
- Active iTBS-DLPFC (Experimental): This active group will receive intermittent theta-burst TMS stimulation.
  Interventions: Device: Active iTBS-DLPFC
- Sham TBS-DLPFC or Sham rTMS-DLPFC (Sham Comparator): Patients in the sham group will receive the same iTBS or rTMS parameter stimulation, performing by a sham coil.
  Interventions: Device: Sham TBS-DLPFC or Sham rTMS-DLPFC

INTERVENTIONS:
Device: Active rTMS-DLPFC — Participants in the rTMS active stimulation group will receive 4-week 10 Hz 120% of RMT to left DLPFC. Left side DLPFC will be targeted by MRI-neuronavigation system. Stimulation will be delivered to the L-DLPFC using a Magstim stimulator.
  Arms: Active rTMS-DLPFC
Device: Active iTBS-DLPFC — Participants in the intermittent TBS(iTBS) active stimulation group will receive 4-week three-pulse 50-Hz bursts administered every 200 milliseconds (at 5 Hz) at an intensity of 80% active motor threshold (MT) to left DLPFC. Left side DLPFC will be targeted by MRI-neuronavigation system. Stimulation will be delivered to the L-DLPFC using a Magstim stimulator.
  Arms: Active iTBS-DLPFC
Device: Sham TBS-DLPFC or Sham rTMS-DLPFC — Half of the patients in the sham group received 4-week the same iTBS parameter stimulation (sham-iTBS), and the other half received the same rTMS parameter stimulation using a sham coil (sham-rTMS), which also improved the blinding process.
  Arms: Sham TBS-DLPFC or Sham rTMS-DLPFC

SUMMARY:
This study evaluates an association between brain-derived neurotrophic factor(BDNF) polymorphisms and the antidepressant efficacy of transcranial magnetic stimulation device in patients with treatment-resistant depression. In a double-blind design, All patients are randomized to three groups, i.e.repetitive transcranial magnetic stimulation treatment, intermittent theta-burst stimulation treatment or sham treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 21 to 70 years of age.
* Diagnosed with the recurrent Major depressive disorder (MDD) and currently having a Major Depressive Episode (MDE)
* Participants failed to respond to at least one adequate antidepressant treatment in their current episode
* Participants have a Clinical Global Impression - Severity score of at least 4 and a total score of at least 18 on the Hamilton Depression Rating Scale (HDRS-17) at both screening and baseline visits ( Day -14 and Day 0)
* Participants must discontinue their antidepressant medications at least for one week ( at least two weeks if Fluoxetine) prior to the TMS intervention and keep antidepressant-free during the study duration.

Exclusion Criteria:

* a lifetime psychiatric history of bipolar disorder, schizophrenia, psychotic disorders, or organic mental disorder including substance abuse and dependence (based on DSM-IV criteria)
* Participants with a lifetime medical history of major systemic illness and clinically significantly abnormal screening examination that might affect safety, study participation, or confound interpretation of study results.
* Participants with a lifetime medical history of neurological disorder records (e.g., stroke, seizure, traumatic brain injury, post brain surgery), brain implants (neurostimulators), cardiac pacemakers
* Women with breastfeeding or pregnancy
* Participants with a current strong suicidal risk (i.e., a score of 4 on item 3 of the HDRS-17)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage change in 17-item Hamilton Depression Rating Scale | Baseline, Week 1, Week 2, Week 3, Week 4(day 20)
  the altered percentage of 17-item Hamilton Depression Rating Scale (range, 0 to 52, with higher scores indicating more depression)

SECONDARY OUTCOMES:
Response rate after 4-week treatment at the end of TMS sessions and three month after. | Baseline, Week 1, Week 2, Week 3, Week 4, week 16 (day 80)
  improvement > 50 % of 17-item Hamilton Depression Rating Scale (range, 0 to 52, with higher scores indicating more depression)
Remission rate after 4-week treatment | Baseline, Week 1, Week 2, Week 3, Week 4, week 16 (day 80)
  17-item Hamilton Depression Rating Scale ≤7 (range, 0 to 52, with higher scores indicating more depression)
Changes in Clinical Global Index | Baseline, Week 1, Week 2, Week 3, Week 4(day 20)
  Clinical Global Index
Changes in depression severity, rated by self-reported | Baseline, Week 1, Week 2, Week 3, Week 4(day 20)
  Depression and Somatic Symptoms Scale, range from 0 to 66 with higher scores indicating more depressive and somatic symptom.
Changes in Young Mania Rating Scale | Baseline, Week 1, Week 2, Week 3, Week 4(day 20)
  Young Mania Rating Scale, range from 0 to 60 with higher scores indicating more severe manic symptoms.
The association between BDNF Polymorphism genotype and the antidepressant efficacy of brain stimulation | Baseline, Week 4(day 20)
  Val/Val, Met/Met, Val/Met genotype and the efficacy after receiving 4-week treatment. The antidepressant efficacy defined by the altered percentage of 17-item Hamilton Depression Rating Scale
The association between the value of baseline brain metabolism and the antidepressant efficacy of brain stimulation | Baseline, Week 4(day 20)
  baseline PET/MRI.The antidepressant efficacy defined by the altered percentage of 17-item Hamilton Depression Rating Scale.
The association between the value of Baseline treatment refractory level and the antidepressant efficacy of brain stimulation | Baseline, Week 4(day 20)
  Maudsley staging method. The antidepressant efficacy defined by the altered percentage of 17-item Hamilton Depression Rating Scale.
The association between the value pf baseline Life event stress scale and the antidepressant efficacy of brain stimulation | Baseline, Week 4(day 20)
  Life event stress scale,range from 0 to 1467 with higher scores indicating more life event stress. The antidepressant efficacy defined by the altered percentage of 17-item Hamilton Depression Rating Scale.
Changes in EEG band before and after brain stimulation | Day 1(pre-RECT, post RECT, post 1st treatment, pre-20th treatment)
  Perform rACC-engaging cognitive task(RECT) before 1-st treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No